CLINICAL TRIAL: NCT03575195
Title: Microbiota Intervention to Change the Response of Parkinson's Disease
Acronym: MICRO-PD
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Conducting an interim analysis
Sponsor: University of California, San Francisco (Other)
Collaborators: Nova Southeastern University (Other); Gateway Institute for Brain Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-22841
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Rifaximin
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 550mg orally
  Arms: Intervention
Other: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
The clinical phenotype of Parkinson's disease (PD) is quite variable, as is the response to and side effects from medications. While many patients respond to carbidopa/levodopa early on, motor fluctuations and dyskinesias can become a problem as the condition progresses, causing significant impairment in function and quality of life. The gut microbiome is of increasing interest in PD, potentially contributing to pathophysiology and clinical phenotype. Furthermore, gut bacteria are capable of metabolizing levodopa, which may decrease its ability to reach the central nervous system and could explain the variable effect seen clinically. Altering the population of drug-metabolizing bacteria could improve the clinical symptoms of PD and the benefit seen with medications. The investigators hypothesize that the gut microbiome in people with PD correlates with their phenotypic characteristics, which can be improved with targeting the microbiome through dietary or therapeutic interventions. The investigators propose a two-part clinical trial. First, a cross-sectional analysis will correlate the microbiome profile with (a) the clinical phenotype of PD and (b) medication response. Second, a randomized, controlled trial, will evaluate the effect of microbiome manipulation on clinical phenotype and medication response. The investigators plan to reduce the level of bacteria through antibiotic use, resetting the potentially disadvantageous microbiome population. Outcomes will include changes in clinical symptoms, alterations in the the microbiome, and changes in serum markers of inflammation. This thorough characterization will broaden our understanding of the gut-brain axis significantly in PD in clinically relevant ways that have yet to be explored.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Stable on levodopa therapy with fluctuations

Exclusion Criteria:

* Chronic gastrointestinal disease
* Recent antibiotic or probiotic therapy
* Pregnant
* Immunocompromised

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS Part III | Two weeks
  The Movement Disorders Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a validated scale that quantifies many of the symptoms and signs of Parkinson's disease. Part III in particular focuses on the motor symptoms of Parkinson's disease through a neurologic exam. The exam is often performed when medications are held for 8-12 hours (the "OFF" state) and again when medications are given and providing therapeutic benefit (the "ON" state), and the difference between scores is calculated. The scale goes from a minimum of 0 to a maximum of 132. There is no specific cutoff, but a higher score indicates a higher severity of symptoms. The trial will examine the change in the MDS-UPDRS Part III both OFF and ON medication after the intervention.
Percent of OFF time according to home motor diaries | Two weeks
  Patients with Parkinson's disease often have times where levodopa is providing therapeutic benefit and times when it is not. "OFF" time indicates the times of day where levodopa therapy is not providing therapeutic benefit. An outcome of the trial will be the change in medication OFF time that the participant experiences at home, according to motor diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Tanner, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No